CLINICAL TRIAL: NCT02975388
Title: A Multi-Center, Open-Label, Two-Part Study to Investigate the Effect of Renal Function and Hemodialysis on the Pharmacokinetics of RO7079901
Brief Title: A Study to Investigate the Effect of Renal Function and Hemodialysis on the Pharmacokinetics (PK) of RO7079901
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NP39380
Record Dates: First submitted 2016-11-24; First posted 2016-11-29 (Estimated); Last update posted 2017-12-11 (Actual); Status verified 2017-12

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency

ARMS (5):
- Label: RO7079901 (Mild) (Part 1) (Experimental): Participants with mild renal impairment (but not undergoing hemodialysis) will be enrolled in this arm. Participants will receive the specified dose of RO7079901.
  Interventions: Drug: RO7079901
- RO7079901 (Moderate) (Part 1) (Experimental): Participants with moderate renal impairment (but not undergoing hemodialysis) will be enrolled in this arm. Participants will receive the specified dose of RO7079901.
  Interventions: Drug: RO7079901
- RO7079901 (Severe) (Part 1) (Experimental): Participants with severe renal impairment (but not undergoing hemodialysis) will be enrolled in this arm. Participants will receive the specified dose of RO7079901.
  Interventions: Drug: RO7079901
- RO7079901 (Normal) (Part 1) (Active Comparator): Control group of participants with normal renal function will be enrolled in this arm. Participants will receive the specified dose of RO7079901.
  Interventions: Drug: RO7079901
- RO7079901 (End-stage) (Part 2) (Experimental): Participants with stable end-stage renal disease undergoing hemodialysis will be enrolled in this arm. Participants will receive the specified dose of RO7079901.
  Interventions: Drug: RO7079901

INTERVENTIONS:
Drug: RO7079901 — Participants will receive a single dose of 1000 milligrams (mg) RO7079901 as a 30-minute intravenous (IV) infusion.

SUMMARY:
This is a multi-center, non-randomized, open-label, two-part study to investigate the effect of renal function and hemodialysis on PK of RO7079901. Part 1 will be conducted in adult male and female participants with stable mild, moderate or severe renal impairment and a control group of participants with normal renal function. Part 2 will be conducted in adult male and female participants with stable end-stage renal disease undergoing hemodialysis.

ELIGIBILITY:
Inclusion Criteria:

- Body Mass Index (BMI) between 18 and 38 kilograms per square-meter (kg/m^2) and body weight of at least 45 kilograms (kg)

Control group participants, Part 1 only:

* Normal renal function based on creatinine clearance greater than or equal to (>=) 90 milliliters per minute (mL/min) at the Screening visit
* Healthy for age-group, as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs, and 12-lead electrocardiogram (ECG)

Participants with renal impairment, Part 1 only:

* Reduced renal function based on estimated creatinine clearance at the Screening visit. Creatinine clearance can be estimated from serum creatinine concentration at the Screening visit using the Cockcroft-Gault equation, or be a historical measured value obtained within the preceding 3 months. Participants with severe, moderate or mild renal impairment must have creatinine clearance of less than or equal to (<=) 29, 30 to 59, or 60 to 89 mL/min, respectively
* Stable renal function. The stability of renal function will be confirmed by two determinations of serum creatinine separated by at least 7 days (one of which can be a historical value within the last 3 months). Renal function will be considered stable if the 2 serum creatinine values differ by <=30 percent (%) of the lower value

Participants with end-stage renal disease in Part 2 only:

* Reduced renal function with a clinical diagnosis of end-stage renal disease requiring renal replacement therapy
* Receiving hemodialysis for more than 3 months at the time of the Screening visit

Exclusion Criteria:

* Recipient of a renal transplant (Part 1 only)
* Presence of renal carcinoma, or acute renal disease caused by infection or drug toxicity
* Nephrotic syndrome (defined as plasma albumin less than [<] 3 grams per deciliter [g/dL] and/or proteinuria greater than [>] 3 grams per day [g/day])
* Hemoglobin concentration <10 g/dL, or <9 g/dL for participants with end-stage renal disease
* Potassium concentration >5.5 millimoles per liter (mmol/L)
* Clinically significant liver disease
* Uncontrolled blood pressure
* Any condition associated with intra-vascular volume depletion
* Any unstable clinically significant disease
* Any other ongoing condition or disease (apart from renal dysfunction), or clinically significant abnormalities in laboratory test results that the investigator considers would render the participant unsuitable for the study, place the participant at undue risk or interfere with the ability of the participant to complete the study
* Major surgery or significant traumatic injury <28 days prior to the first administration (excluding biopsies), or anticipation of the need for major surgery during study treatment
* Recent history of alcoholism, drug abuse, or addiction within the last year prior to screening
* Positive test at Screening of any of the following: Hepatitis A, Hepatitis B, Hepatitis C, or human immunodeficiency virus (HIV)
* Clinically significant change in disease status as judged by the investigator, or any major illness within the 4 weeks prior to the Screening visit, or febrile illness within 14 days prior to the Screening visit
* Use of prohibited medications, or alteration to a concomitant medication treatment regimen considered relevant by the investigator within 14 days before the Screening visit
* Known history of clinically significant hypersensitivity or severe allergic reaction to any drug, in particular antibiotics (e.g., cephalosporins, penicillins, carbapenems, or monobactams)
* Participation in another clinical study with an investigational drug or device within the 1 month preceding the Screening vist
* Donation or loss of over 500 milliliters (mL) of blood within the 3 months before the Screening visit

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-12-20 (Actual); Primary Completion 2017-07-06 (Actual); Study Completion 2017-07-06 (Actual)

PRIMARY OUTCOMES:
Total Body Clearance (CL) of RO7079901 Using Plasma Concentration Data | Blood: Part 1 - Predose (-1 to 0 hour [hr]), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Volume of Distribution of the Central Compartment (Vc) of RO7079901 Using Plasma Concentration Data | Blood: Part 1 - Predose (-1 to 0 hr), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Total Volume of Distribution (Vz) of RO7079901 Using Plasma Concentration Data | Blood: Part 1 - Predose (-1 to 0 hr), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Volume of Distribution at Steady-State (Vss) of RO7079901 Using Plasma Concentration Data | Blood: Part 1 - Predose (-1 to 0 hr), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Renal Clearance (CLr) of RO7079901 | Urine: Part 1 - 0-4, 4-8, 8-12, 12-24 hr postdose; Part 2 - 0-12 hr postdose ( infusion length: 0.5 hr)
Part 2: Dialysis Clearance (CLd) of RO7079901 | Dialyzer input, output blood and dialyzer fluid: 1.5 hours postdose (start of hemodialysis); 2.5, 3.5, 4.5 hours postdose (end of hemodialysis) (infusion length: 0.5 hr)
Measured Creatinine Clearance (mCLcr) | Blood and Urine: Day -1 ( over the 24-hr period predose corresponding to time of micturition), Day 1 ( Part 1)
Estimated Creatinine Clearance Using the Cockcroft and Gault Formula (eCLcr[CG]) | Blood and Urine: Day -1 (over the 24-hr period predose corresponding to time of micturition), Day 1 (Part 1)
Estimated Creatinine Clearance Using the Modified Jelliffe Formula (eCLcr[Jelliffe]) | Blood and Urine: Day -1 (over the 24-hr period predose corresponding to time of micturition), Day 1 (Part 1)
Estimated Glomerular Filtration Rate (eGFR) Using the Modification of Diet in Renal Disease (MDRD) Formula (eGFR[MDRD]) | Blood and Urine: Day -1 (over the 24-hr period predose corresponding to time of micturition), Day 1 (Part 1)
eGFR Using the Chronic Kidney Disease Epidemiology (CKD-EPI) Formula (eGFR[CKD-EPI]) | Blood and Urine: Day -1 (over the 24-hr period predose corresponding to time of micturition), Day 1 (Part 1)

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve From Time 0 to infinity (AUC0-inf) of RO7079901 | Blood: Part 1 - Predose (-1 to 0 hr), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Maximum Plasma Concentration (Cmax) of RO7079901 | Blood: Part 1 - Predose (-1 to 0 hr), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Time to Reach Cmax (tmax) of RO7079901 | Blood: Part 1 - Predose (-1 to 0 hr), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Terminal Elimination Half-life (t1/2) of RO7079901 | Blood: Part 1 - Predose (-1 to 0 hr), 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, and 24 hr postdose; Part 2 - Predose (-1 to 0 hr), 0.5, 1, 1.5 (start of hemodialysis), 4.5 (end of hemodialysis), 8, 12, and 24 hr postdose (infusion length: 0.5 hr)
Cumulative Amount Excreted in Urine (Ae) of RO7079901 | Urine: Part 1 - 0-4, 4-8, 8-12, 12-24 hr postdose; Part 2 - 0-12 hr postdose (infusion length: 0.5 hr)
Fraction Excreted in Urine (Fe) of RO7079901 | Blood:Predose (-1 to 0hr), 0.5, 1, 1.5, 8, 12, 24 hr postdose(Parts 1 and 2); 2, 3, 4, 6 hr postdose(Part 1); 4.5 hr postdose(end of hemodialysis)(Part 2); Urine:0-4, 4-8, 8-12, 12-24 hr postdose(Part 1); 0-12 hr postdose(Part 2)(infusion length: 0.5 hr)
Percentage of Participants with Adverse Events (AEs) | Baseline up to end of the study (up to approximately 7 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-LaRoche
Locations (5):
- United States (5):
  - Clinical Pharmacology of Miami, Inc., Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota
  - Prism Clinical Research, Saint Paul, Minnesota
  - New Orleans Center for Clinical Research, Knoxville, Tennessee